CLINICAL TRIAL: NCT02312934
Title: Nicotinic Treatment of Post-Chemotherapy Subjective Cognitive Impairment: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Paul Newhouse, Professor of Psychiatry, Pharmacology, and Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 141584
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Chemo Brain; Chemotherapy-related Cognitive Impairment; Chemo Fog; Breast Cancer; Chemobrain
Keywords: Chemo brain; Chemotherapy-related cognitive impairment; CRCI; Breast cancer; Chemo fog; Nicotine; Transdermal nicotine
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Breast Neoplasms | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdermal Nicotine (Experimental): Nicotine will be delivered by a transdermal patch delivery system for topical application. Each patch will contain approximately 1.75mg nicotine/cm2, and releases 7, and 14mg of nicotine, respectively, over 24 hours. Patches will be applied for 16 hours per day. Participants will be titrated over the course of the 6-week treatment period in order to avoid initial side effects as follows:
  Week 1: ½ 7 mg patch per day, Week 2: 7 mg patch per day, Weeks 3-4: ¾ 14 mg patch per day, Weeks 5-6: 14 mg per day, Weeks 7-8: Treatment withdrawal
  Interventions: Drug: Transdermal nicotine
- Placebo (Placebo Comparator): Matching transdermal placebo patches will be used. Participants will follow the same titration schedule as the transdermal nicotine arm.
  Week 1: ½ 7 mg patch per day, Week 2: 7 mg patch per day, Weeks 3-4: ¾ 14 mg patch per day, Weeks 5-6: 14 mg per day, Weeks 7-8: Treatment withdrawal
  Interventions: Other: Placebo Transdermal Patch

INTERVENTIONS:
Drug: Transdermal nicotine — Nicotine patches are currently FDA approved for smoking cessation. Nicotine has effects that have been well studied for many years. Studies have shown that nicotine by itself does not appear by itself to be cancer causing. The use of the nicotine patch is not expected to increase risk of breast cancer recurrence.
  Arms: Transdermal Nicotine
Other: Placebo Transdermal Patch — Matching transdermal placebo patches will be used. Participants will follow the same titration schedule as the transdermal nicotine arm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the use of a nicotine patch as a treatment for problems with attention, learning and memory in breast cancer patients who are 1-5 years post chemotherapy.

DETAILED DESCRIPTION:
Studies have suggested that chemotherapy treatment for breast cancer may change the way the brain functions. As a result, patients who receive chemotherapy for breast cancer may experience problems with their attention, learning, and memory that they did not have before receiving chemotherapy. The investigators have found that nicotine treatment can help other types of patients with similar difficulties with attention, learning, and memory. Nicotine is a naturally occurring substance found in tobacco and is known to interact with nerve cells in the brain that are important for functions like learning and memory, and has been studied in a number of disorders. This study is designed to test whether nicotine treatment is helpful for learning and memory problems after chemotherapy for breast cancer.

This study will be a randomized, placebo-controlled pilot study to evaluate the effect of transdermal nicotine to 1) reduce subjective complaints and 2) enhance cognitive performance on laboratory measures of cognitive performance in breast cancer patients with persistent chemotherapy-related cognitive impairment (CRCI), a condition also known as "chemo brain." Participants will be randomized to either placebo or active compound (50/50) for the 6-week treatment portion of the study. Participants will be assessed before, during, and at the end of treatment. At the end of the 8-week study, participants will have the option to take part in the open-label portion of the study for an additional 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All participants will:

  1. Be between 35 and 80 years of age,
  2. Have been diagnosed with noninvasive or invasive (Stage 1, 2, or 3A) breast cancer,
  3. Have undergone treatment with systemic chemotherapy within the last 1-5 years,
  4. Endorse persistent CRCI subjective complaints,
  5. Be non-smokers (no nicotine use within the last 5 years),
  6. Have no active cardiac, neurologic, or psychiatric illness, and
  7. Fluent in and able to read English.

Exclusion Criteria:

* Participants will be excluded for:

  1. Any active neurologic and/or psychiatric disease, history of significant head trauma followed by persistent neurologic deficits, or known structural brain abnormalities,
  2. Current major depression or another major psychiatric disorder as described in DSM-5 (use of CNS active medications (e.g. antidepressants) will be permitted, provided dosing has been stable for at least 3 months),
  3. Any history of alcohol or substance abuse or dependence within the past 2 years (DSM-5 criteria),
  4. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol including:
* History of myocardial infarction in the past year or unstable, severe cardiovascular disease including angina or CHF with symptoms at rest, or clinically significant abnormalities on the ECG
* Clinically significant and/or unstable pulmonary, gastrointestinal, hepatic, or renal disease
* Insulin-requiring diabetes or uncontrolled diabetes mellitus,
* Uncontrolled hypertension (systolic BP> 170 or diastolic BP> 100), 5. Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening, and 6. Use of any drugs with pro-cholinergic properties (e.g. donepezil).

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Newhouse, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Center for Cognitive Medicine at Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through Vanderbilt University-affiliated clinics and the greater Nashville, TN community.
Pre-assignment Details: Of the 106 people pre-screened for the study, 37 attended the initial screening visit. Twenty-two participants met entry criteria and were randomized. Participants that were not randomized were excluded from the study because they did not meet inclusion/exclusion criteria.
Groups:
- Transdermal Nicotine: Nicotine will be delivered by a transdermal patch delivery system for topical application. Each patch will contain approximately 1.75mg nicotine/cm2, and releases 7, and 14mg of nicotine, respectively, over 24 hours. Patches will be applied for 16 hours per day. Participants will be titrated over the course of the 6-week treatment period in order to avoid initial side effects as follows:
  Week 1: ½ 7 mg patch per day, Week 2: 7 mg patch per day, Weeks 3-4: ¾ 14 mg patch per day, Weeks 5-6: 14 mg per day, Weeks 7-8: Treatment withdrawal
  Transdermal nicotine: Nicotine patches are currently FDA approved for smoking cessation. Nicotine has effects that have been well studied for many years. Studies have shown that nicotine by itself does not appear by itself to be cancer causing. The use of the nicotine patch is not expected to increase risk of breast cancer recurrence.
- Placebo: Matching transdermal placebo patches will be used. Participants will follow the same titration schedule as the transdermal nicotine arm.
  Week 1: ½ 7 mg patch per day, Week 2: 7 mg patch per day, Weeks 3-4: ¾ 14 mg patch per day, Weeks 5-6: 14 mg per day, Weeks 7-8: Treatment withdrawal
  Placebo Transdermal Patch
Period: Overall Study
Arm/Group | Transdermal Nicotine | Placebo
Started | 11 | 11
Completed (Number Completed) | 9 | 11
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal Nicotine | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.00 (11.58) | 52.55 (7.66) | 54.27 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 10 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 25
Cancer Type [Count of Participants; unit: Participants]
  Breast Cancer | 8 | 10 | 18
  Non-Hodgekin's Lymphoma | 2 | 0 | 2
  Ovarian Cancer | 0 | 1 | 1
  Colon Cancer | 1 | 0 | 1
Cancer Stage [Count of Participants; unit: Participants]
  Stage I | 3 | 5 | 8
  Stage II | 3 | 4 | 7
  Stage III | 4 | 1 | 5
  Stage IV | 1 | 1 | 2
Cancer Treatment Received [Number; unit: participants]
  Chemotherapy | 11 | 11 | 22
  Surgery | 10 | 11 | 21
  Radiation | 5 | 7 | 12
Current Endocrine Therapy [Count of Participants; unit: Participants]
  Yes | 6 | 7 | 13
  No | 5 | 4 | 9
Post-Menopausal Status [Count of Participants; unit: Participants]
  Pre-Menopausal | 5 | 6 | 11
  Post-Menopausal | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) PCI Scale
Description: The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) scale will be used to monitor change in CRCI subjective complaints.
  This instrument has been used to monitor change in CRCI subjective complaints in previous studies and demonstrates good internal consistency, test-retest reliability, and discriminant and convergent validity. Specifically, the PCI subscale was used as the primary outcome measure.
  The FACT-Cog PCI consists of 20 items and has a minimum score of 0 and total possible score of 72. Higher scores indicate better cognitive functioning.
  The PCI evaluates memory, concentration, mental acuity, verbal fluency, functional interference, and multitasking ability.
  Visit 3 is the 3-week visit, Visit 4 is the 6-week visit, and Visit 5 is the 8-week visit.
  Change scores were calculated as follow
Time Frame: Baseline to 8-Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  Visit 3 PCI Change from Baseline Score (3-Weeks) | 7.00 (12.01) | 11.55 (9.59)
  Visit 4 PCI Change from Baseline Score (6-Weeks) | 16.80 (15.47) | 16.64 (7.58)
  Visit 5 PCI Change from Baseline Score (8-Weeks) | 11.20 (14.40) | 16.55 (10.40)
Statistical Analysis 1: Comparison: Transdermal Nicotine vs Placebo; For the Primary Aim (Specific Aim 1), a mixed-models repeated measures ANOVA was used to assess the interaction of treatment group (nicotine, placebo) with time (Visit), using change from baseline PCI FACT-Cog score (Visit 3, Visit 4, and Visit 5) as the dependent measure; Test type: Other; p = 0.41, Mixed Models Analysis — All pairwise comparisons were Sidak corrected for multiple comparisons at the p < 0.05 level; Degrees of freedom were corrected using Greenhouse-Geisser estimates of sphericity (ε = 0.72)

2. Secondary Outcome: Conners Continuous Performance Test
Description: The secondary outcome measure was the computerized Conners Continuous Performance Test (CPT), which measures sustained attention and vigilance. Participants see a series of letters appearing one at a time on a computer screen and they press a button for every letter that appears on the screen, except for "X". Lower scores indicate better performance.
  Scores on the CPT are calculated using the each participant's performance on the task (defined as reaction time (in ms) standard error/interstimulus interval). Change scores from baseline are then calculated. A decrease in CPT score = improvement.
  *This is not a clinical measure. This is a research measure of reaction time variability and therefore there is no clinical interpretation and no defined score range.*
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Placebo: Matching transdermal placebo patches will be used. Participants will follow the same titration schedule as the transdermal nicotine arm.
  Week 1: ½ 7 mg patch per day, Week 2: 7 mg patch per day, Weeks 3-4: ¾ 14 mg patch per day, Weeks 5-6: 14 mg per day, Weeks 7-8: Treatment withdrawal
  Placebo Transdermal Patch: Matching transdermal placebo patches will be used. Participants will follow the same titration schedule as the transdermal nicotine arm.
Arm/Group | Transdermal Nicotine | Placebo
Number analyzed (Participants) | 11 | 11
ms
  Visit 3 CPT Change from Baseline Score (3-Weeks) | 0.0127 (0.11705) | -0.0318 (0.1256)
  Visit 4 CPT Change from Baseline Score (6-Weeks) | 0.01 (0.17205) | -0.0355 (0.12242)
  Visit 5 CPT Change from Baseline Score (8-Weeks) | -0.0185 (0.19357) | -0.0236 (0.14009)
Statistical Analysis 1: Comparison: Transdermal Nicotine vs Placebo; For the Secondary Aim (Specific Aim 2), a mixed-models repeated measures ANOVA was used to assess the interaction of treatment group (nicotine, placebo) with time (Visit), using change from baseline CPT Scores (Visit 3, Visit 4, and Visit 5) as the dependent measure; Test type: Other; p = 0.79, Mixed Models Analysis — All pairwise comparisons were Sidak corrected for multiple comparisons at the p < 0.05 level; Degrees of freedom were corrected using Greenhouse-Geisser estimates of sphericity (ε = 0.72)

ADVERSE EVENTS:
Time Frame: 8-Weeks
Description: Adverse events were recorded and categorized by body system, event type, attribution, frequency, severity, and course. AEs were assessed across all double-blind study visits and categorized according to body system for all participants who received at least one dose of patches (nicotine n = 12, placebo n = 13).
Arm/Group | Transdermal Nicotine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 7/11 | 8/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Nicotine (N=11) | Placebo (N=11)
Skin Irritation (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 3 (3) — Nausea
Neurologic (General disorders) | 2 (2) | 2 (2) — Dizziness
Mood (General disorders) | 0 (0) | 1 (1) — Irritability
Insomnia (General disorders) | 0 (0) | 1 (1) — Insomnia

LIMITATIONS AND CAVEATS:
Small sample size numbers; treatment duration of 6-weeks may not have been enough time to distinguish between a drug and placebo response; 14mg may not have been a sufficient dose to fully test this hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT02312934/Prot_SAP_000.pdf